CLINICAL TRIAL: NCT05998330
Title: LiverPAL: A Randomized Trial of Inpatient Palliative Care for Patients With Advanced Liver Disease
Brief Title: LiverPAL: A Trial of Inpatient Palliative Care for Patients With Advanced Liver Disease
Acronym: LiverPAL
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Nneka nnaoke Ufere, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023P001894; 80736 (Other Grant/Funding Number: Robert Wood Johnson Foundation); 242379 (Other Grant/Funding Number: Cambia Health Foundation); 243432 (Other Grant/Funding Number: American Association for the Study of Liver Diseases); 236965 (Other Grant/Funding Number: Massachusetts General Hospital Executive Committee on Researrch)
Record Dates: First submitted 2023-08-11; First posted 2023-08-18 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Liver Disease Chronic; End Stage Liver DIsease; Cirrhosis; Cirrhosis, Liver; Advanced Cirrhosis
MeSH Terms: conditions — End Stage Liver Disease; Fibrosis; Liver Cirrhosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Usual Hepatology Care (No Intervention): Usual hepatology care
- Usual Hepatology Care with Early Palliative Care (Experimental): Usual hepatology care with early palliative care
  Interventions: Behavioral: LiverPAL

INTERVENTIONS:
Behavioral: LiverPAL — The intervention include integrating early palliative care with usual hepatology care to evaluate and treat patients' symptoms, enhance their illness and prognostic understanding, support their coping, and coordinate their serious illness, transitional, and end-of-life care.
  Arms: Usual Hepatology Care with Early Palliative Care

SUMMARY:
The goal of this clinical trial is to evaluate whether early integration of palliative care in the care of hospitalized patients with advanced liver disease (AdvLD) can improve patients' quality of life, physical symptoms, mood, and serious illness communication. Palliative care is a medical specialty focused on lessening (or "palliating") symptoms and assisting in coping with serious illness.

DETAILED DESCRIPTION:
The main purpose of this study is to compare two types of care - usual hepatology care and usual hepatology care with early involvement of palliative care clinicians to see which is better for improving the experience of hospitalized patients with advanced liver disease (AdvLD).

The investigators aim to find out whether introducing hospitalized patients with AdvLD to the palliative care team that specializes in symptom management can improve the quality of life and physical and psychological symptoms that patients and families experience during their hospitalizations as well as enhance the quality of patients' end of life care.

ELIGIBILITY:
Patient Inclusion Criteria:

1. Hospitalized patient with a diagnosis of advanced liver disease, defined as cirrhosis with one of the following (new or ongoing) within the prior six months from date of consent:

   * Ascites (requiring diuretics or serial large volume paracenteses)
   * Spontaneous bacterial peritonitis
   * Hepatic hydrothorax (requiring diuretics)
   * Variceal bleed (with one or more occurrences)
   * Overt hepatic encephalopathy (requiring medications)
2. Ability to comprehend English

Patient Exclusion Criteria:

1. Prior history of liver transplantation
2. Have uncontrolled hepatic encephalopathy, cognitive impairment, psychiatric disorder or other comorbid condition which the primary medical, hepatology, and/or transplant surgery teams believes prohibits the ability to provide informed consent
3. Current or recent (within 5 years of receiving curative cancer treatment) history of extrahepatic malignancy (excluding non-melanoma skin cancer)
4. Presence of hepatocellular carcinoma beyond Milan criteria
5. Are already receiving hospice care
6. Receive a score of <10 on the Simplified Animal Naming Test

Caregiver Inclusion Criteria

1. Adult caregiver (≥ 18 years of age)
2. A relative or friend identified by the patient upon whom the patient relies for help and who likely is to be present in-person during hospitalizations or clinic appointments, or willing to participate by phone
3. Ability to comprehend English and can complete questionnaires

Caregiver Exclusion Criteria

1. Inability to comprehend English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-09-20 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Patient Quality of Life (Functional Assessment of Chronic Illness Therapy - Palliative Care, FACIT-Pal) up t0 4 weeks | Up to 4 weeks
  Compare patient quality of life (FACIT-Pal) scores up to 4 weeks adjusting for baseline quality of life scores between the study arms. Score range 0-184 with higher scores indicating better quality of life.

SECONDARY OUTCOMES:
Patient FACIT-Pal Score longitudinally between study arms | Up to 6 months
  Compare patient quality of life (FACIT-Pal) scores longitudinally between the study arms. Score range 0-184 with higher scores indicating better quality of life.
Patient Symptom Burden (revised Edmonton Symptom Assessment Scale, ESAS-r) | Up to 6 months
  Compare patient symptom burden scores (ESAS-r) between the study arms. Score range 0-100 with higher scores indicating higher symptom burden.
Patient Depression Symptoms (Hospital Anxiety and Depression Scale, HADS-D) | Up to 6 months
  Compare patient depression symptoms (HADS-D) between the study arms. Score range 0-21 with higher scores indicating higher depression symptoms.
Patient Anxiety Symptoms (Hospital Anxiety and Depression Scale, HADS-A) | Up to 6 months
  Compare patient anxiety symptoms (HADS-A) between study arms. Score range 0-21 with higher scores indicating higher anxiety symptoms.
Patient End-of-Life (EOL) Care Communication with Clinicians | Final assessment prior to patient death or at 6 months
  "Has [participant] talked with [participant's] doctor about the kind of medical care [participant] would want if [participant] were very sick or near the end of life?"
Documentation of Patient End-of-Life (EOL) Care Preferences | After patient death, up to 60 months
  Compare documentation of EOL care preferences in the electronic health record between study arms since baseline.

OTHER OUTCOMES:
Patient End-of-Life (EOL) Care | Within 30 days of patient death
  Compare rate of receipt of intensive EOL care (renal replacement therapy, mechanical ventilation, and/or cardiopulmonary resuscitation or death in the intensive care unit) between study arms.
Caregiver Quality of Life (PROMIS-29+2) | Up to 6 months
  Compare caregiver quality of life (PROMIS-29+2) between study arms. Scores range 4-20 for raw items and 2-10 for cognitive function, with a higher score represents more of the concept being measured. Raw scores are translated into standardized T-scores.
Caregiver Depression Symptoms (Hospital Anxiety and Depression Scale, HADS-D) | Up to 6 months
  Compare caregiver depression symptoms (HADS-D) between study arms. Score range 0-21 with higher scores indicating higher depression symptoms.
Caregiver Anxiety Symptoms (Hospital Anxiety and Depression Scale, HADS-A) between study arms. | Up to 6 months
  Compare caregiver anxiety symptoms (HADS-A) between study arms. Score range 0-21 with higher scores indicating higher anxiety symptoms.
Caregiver Burden (Zarit Burden Index 12, ZBI-12) | Up to 6 months
  Compare caregiver burden scores (ZBI-12) between study arms. Score range 0-48 with higher scores indicating higher caregiver burden.
Receipt of goal-concordant end-of-life care - patient wishes followed | At least 1 month after patient death, up to 3 months
  Bereaved caregivers will be asked "In [participant's] opinion, to what extent were [the patient's] wishes followed in the medical care received in the last month of life?" Receipt of goal-concordant end-of-life care - patient wishes followed will be defined as care that "followed patients' wishes a great deal."
Quality of Life Near Death (QOD) | After patient death, up to 60 months
  Bereaved caregivers will be asked "Just prior to the death of [the patient] (eg, his/her last week; when last seen), how would [participant] rate [the patient's] level of…" (1) "psychological distress?" (0 = none; 10 = extremely upset); (2) "physical distress?" (0 = none; 10 = extremely distressed); and (3) "overall quality of life in the last week of life/death?" (0 = worst possible; 10 = best possible). Ratings for these three items will be averaged (with reverse coding for the psychological and physical distress items). Scores range 0-10 with higher composite scores representing better QOD.
Prolonged Grief Disorder (PG-13-R) | At least 12 months after patient death, up to 60 months
  Compare rates of prolonged grief disorder (PG-13-R) among bereaved caregivers between study arms. Score range 10-50 for symptom items with higher scores indicating worsening symptoms.
Healthcare Utilization at End-of-Life - Hospice | After patient death, up to 60 months
  Compare rates of hospice utilization (yes/no) between study arms.
Healthcare Utilization at End-of-Life - Hospice length of stay | After patient death, up to 60 months
  Compare number of days in hospice for patients admitted to hospice between study arms.
Healthcare Utilization - Days alive and out of the hospital | Up to 6 months
  Compare days alive and out of the hospital at 6 months (180 days) after randomization
Healthcare Utilization - liver transplantation | Up to 60 months
  Compare rates of liver transplantation (yes/no) between study arms
Patient Coping (Brief COPE) | Up to 6 months
  Compare patient coping using the Brief Cope questionnaire between study arms. We will administer 14 items of the Brief COPE comprising seven subscales (active coping, use of emotional support, positive reframing, acceptance, behavioral disengagement, denial, and self-blame). Higher scores on each subscale indicate more use of that particular coping strategy.
Caregiver Coping (Brief COPE) | Up to 6 months
  Compare caregiver coping using the Brief Cope questionnaire between study arms. We will administer 14 items of the Brief COPE comprising seven subscales (active coping, use of emotional support, positive reframing, acceptance, behavioral disengagement, denial, and self-blame). Higher scores on each subscale indicate more use of that particular coping strategy.
Patient Feeling Heard and Understood Scale | Up to 6 months
  We will use the validated 4-item scale "Feeling Heard and Understood" as a self-reported measure capturing seriously ill patients' global assessment of their health care quality in the hospital environment. Response options range from 0 (not at all true) to 4 (completely true) for a score range of 0-16.
Caregiver Feeling Heard and Understood Scale | Up to 6 months
  We will use the validated 4-item scale "Feeling Heard and Understood" as a self-reported measure capturing seriously ill patients' caregivers' global assessment of their loved one's health care quality in the hospital environment. Response options range from 0 (not at all true) to 4 (completely true) for a score range of 0-16.
Patient End-of-Life (EOL) Care Communication with Caregivers | Final assessment prior to patient death or at 6 months
  "Has [participant] talked with [participant's] family or friends about the kind of medical care [participant] would want if [participant] were very sick or near the end of life?"
Patient Quality of Life (PROMIS-29+2) | Up to 6 months
  Compare patient quality of life (PROMIS-29+2) scores between study arms. Scores range 4-20 for raw items and 2-10 for cognitive function, with a higher score represents more of the concept being measured. Raw scores are translated into standardized T-scores.

CONTACTS AND LOCATIONS:
Overall Officials: Nneka Ufere, MD MSCE, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No